CLINICAL TRIAL: NCT01194375
Title: A Dose-Ranging Study Evaluating the Safety and Efficacy of IDP-107 in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-IDP-107-P2-02
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Low Strength IDP-107 (Experimental)
  Interventions: Drug: Low Strength IDP-107
- High Strength IDP-107 (Experimental)
  Interventions: Drug: High Strength IDP-107
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Strength IDP-107 — Once a day for 16 weeks
  Arms: Low Strength IDP-107
Drug: High Strength IDP-107 — Once a day for 16 weeks
  Arms: High Strength IDP-107
Drug: Placebo — Once a day for 16 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of IDP-107 versus placebo in treating patients with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Presence of acne vulgaris on the face and neck/trunk
* Presence of inflammatory and non-inflammatory lesions on the face

Exclusion Criteria:

* Presence of any skin condition on the face that could interfere with clinical evaluations
* Use of any systemic antibiotics or corticosteroids within 4 weeks prior to the Baseline visit
* Use of any systemic retinoids, such as isotretinoin, within 3 months prior to the Baseline visit
* Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of inflammatory lesions | Baseline and 22 weeks
Percent of patients who achieve success for the acne global severity score | Baseline and 22 weeks

SECONDARY OUTCOMES:
Change from baseline in the number of non-inflammatory lesions | Baseline and 22 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Dermatology Specialists, Inc., Oceanside, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - FXM Research Corp., Miami, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Pedia Research LLC, Owensboro, Kentucky
  - ActivMed Practices and Research, Inc., Haverhill, Massachusetts
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Oregon Dermatology and Research Center, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - South Valley Dermatology, West Jordan, Utah
  - Premier Clinical Research, Spokane, Washington
- Canada (3):
  - Ultranova Skincare, Barrie, Ontario
  - The Centre for Dermatology and Cosmetic Surgery, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario